CLINICAL TRIAL: NCT05816564
Title: Optimizing Attentional Bias Modification for Depression: Does Mindfulness Help?
Brief Title: Optimizing Attentional Bias Modification
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Tyler (Other)
Collaborators: Psi Chi (Other); Sarah Sass, PhD (Unknown)
Responsible Party: Principal Investigator, Bridget Kennedy, Doctoral Research Assistant, University of Texas at Tyler
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-FY2021-51
Record Dates: First submitted 2023-02-03; First posted 2023-04-18 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Depression
Keywords: Attention Bias; Mindfulness
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to positive attention training or "sham" attention training but will both receive mindfulness exercises.
Who Masked: Participant
Masking Description: Participants will be debriefed after study but are not specifically told that they were recruited due to reported depression symptoms.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): This is group that will receive the attention bias modification intervention that is programmed to train attention to positive stimuli 100% of the time. Both groups will receive the preceding 3-day brief mindfulness training.
  Interventions: Behavioral: Attention Bias Modification (ABM) for depression
- Placebo/Control Group (Placebo Comparator): This is group that will receive the "sham" attention bias modification intervention that is programmed to train attention to positive stimuli 50% of the time. Both groups will receive the preceding 3-day brief mindfulness training.
  Interventions: Behavioral: Sham Attention Bias Modification (ABM)

INTERVENTIONS:
Behavioral: Attention Bias Modification (ABM) for depression — Both groups will be asked to engage in mindfulness activities but only one group will receive the train-positive ABM task. The control group will receive a "sham" task that is not programmed to train attention towards positive stimuli.
  Arms: Experimental Group
Behavioral: Sham Attention Bias Modification (ABM) — The sham intervention will be given to the control group (but they will still receive mindfulness exercises).
  Arms: Placebo/Control Group

SUMMARY:
Depression has been associated with an attention bias towards negative information. Attention bias modification (ABM) interventions explore potential benefits of training attention away from negative or threatening information and towards neutral or positive information. The goal of this study is to examine the effectiveness of an ABM intervention that includes a preceding mindfulness training among a sample of individuals who self-reported mild-to-moderately depression symptoms. The main question this study aims to answer is:

• Do individuals who participate in an ABM intervention have a greater reduction in attention bias towards negative information and depressive symptoms when compared to a control group? Participants will be asked to participate in 3 days of brief mindfulness training exercises preceding an ABM intervention session that lasts 1.5 to 2 hours while wearing electroencephalography (EEG) equipment.

Researchers will compare the ABM intervention group to a "sham" intervention group to see if the ABM intervention reduces negative attention bias above and beyond brief mindfulness training.

DETAILED DESCRIPTION:
Approximately 50 participants who have self-reported mild-to-moderate levels of depression will be invited to participate in the study. They will be asked to participate over the course of 3 days. On the first day, informed consent will be reviewed, the participant will be asked a series of survey questions and asked to begin the first mindfulness exercise. On the second day, the participant will be asked to complete a second mindfulness exercise on their own. On the third day, the participant will be asked to complete a final mindfulness exercise and then to participate in an ABM intervention session while wearing EEG equipment to monitor brain waveforms and extract event-related potentials (ERPs).

The mindfulness activities used for this study were developed for individuals with depression symptoms. The initial activity will consist of introduction to mindfulness with a brief breathing activity developed specifically for individuals suffering from depression symptoms. Participants will complete the first mindfulness activity 2 days prior to their ABM session, the second activity the day before, and refresher activity immediately preceding their ABM intervention. During the ABM intervention session, participants will complete a pre- and post-intervention dot-probe task (DPT) to assess for the presence of attention bias before and after the intervention. The pre- and post-tasks will consist of trials displaying a fixation cross for 500 ms followed by two faces (happy or sad displayed with neutral) on the left and right side of visual space for 2000 ms. These images are selected from the racially diverse affective expression (RADIATE) face stimulus set and randomized. Once the faces are displayed, after a probe, single asterisk or double asterisks will appear in the same location as one of the faces. Probes will replace an emotional or neutral face with equal frequency. Participants will respond to the probe by indicating the number of asterisks they saw using a designated key. The task will consist of 192 trials (two blocks of 96 trials) with 12 pairs of sad and neutral images and 12 pairs of happy and neutral images randomly presented eight times. Stimuli used in pre- and post-tasks are different from stimuli used during training. Emotional stimuli will be matched on valence and arousal in the two task sets. ABM intervention consists of paired positive and negative images and faces. Twenty-two images are presented in nine blocks for a total of 198 trials. A fixation cross is presented in the middle of the screen for 1,500 ms followed by a positive and negative image pair for 4,000 ms. Each type of stimulus will appear with equal probability and pairings are randomized. For the experimental group, probes single or double asterisks will follow the positive stimulus 100% of the time. For the control group, the probe will follow the positive stimulus 50% of the time. Participants will indicate how many asterisks they saw using the indicated key. Participants will be offered breaks after every two blocks to reduce fatigue.

It is expected that individuals who participated in the ABM intervention will demonstrate a more prominent decrease in a negative AB and reduction of depression symptoms when compared to the "sham" group. Outcome measures of this project include reaction time data from ABM intervention task, ERP data from EEG data, and self-report data collected at the beginning and end of the study. Self-report measures used to assess for depression symptoms include the MASQ and Patient Health Questionnaire 9-item (PHQ-9). The PHQ-9 a criteria-based measure used to help diagnose depressive disorders. It was found to be a reliable and valid measure of depression severity and includes a specific item about trouble concentrating. A 4-week follow-up survey with the PHQ-9 will also be sent to participants to assess for any symptom changes at that time. Reaction time (RT) will be used to assess attention bias with faster RT to probes following stimuli with emotion interpreted as attention bias towards that emotion. ERP measures are considered objective; measuring the time course of attention and are expected to support decreased AB towards negative information.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Report of mild-to-moderate levels of depression symptoms.
* Must be able to read and understand English.

Exclusion Criteria:

* Under the age of 18 years old.
* Diagnosed with ADHD.
* Diagnosed with dyslexia.
* Diagnosed with multiple sclerosis.
* Diagnosed with a seizure disorder/epilepsy.
* History of a traumatic brain injury.
* Currently pregnant.
* Unable to read and understand English.
* Difficulty seeing and hearing instructions on a computer.
* Endorsement of current substance abuse problem.
* Having a history of electro-shock therapy.
* Reporting having a medication change in the previous 3-months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Amplitude changes (in microvolts) for scalp-recorded event-related potential (ERP) data. | Changes in ERP amplitudes from the baseline attention task to the final attention task on day 3 of the study.
  ERP data will be captured using Brain Vision software and BrainVision actiCHamp 32channel EEG system. ERP measures are considered objective; measuring the time course of attention and are expected to support decreased AB towards negative information (specifically the P300 and N2pc components).
Reaction Time (RT) | Changes in RT from the baseline attention task to the final attention task on day 3 of the study.
  Reaction time will be collected and used via E-Prime software with a Chronos button box. Reaction time (RT) data is the primary behavioral data used to assess attention bias in ABM research. In the present study, RT will be used to assess attention bias with faster RT to probes following stimuli with emotion interpreted as attention bias.
Patient Health Questionnaire- 9-item | Change from baseline depression symptoms (day 1 of study) to immediately after the 3-day intervention.
  Patient Health Questionnaire- 9-item (PHQ-9) is a self-report assessment used to measure depression symptoms and their severity. Higher scores on the PHQ-9 indicate higher levels of depression symptoms.
Patient Health Questionnaire- 9-item | Change from baseline depression symptoms (day 1 of study) to 4-weeks post-intervention.
  Patient Health Questionnaire- 9-item (PHQ-9) is a self-report assessment used to measure depression symptoms and their severity. Higher scores on the PHQ-9 indicate higher levels of depression symptoms.
Mood and Anxiety Symptom Questionnaire-Anhedonic Depression Subscale | Change from baseline anhedonic depression symptoms (day 1 of study) to immediately after the 3-day intervention.
  The Mood and Anxiety Symptom Questionnaire-Anhedonic Depression Subscale (MASQ-AD8) is a self-report assessment used to measure symptoms of anhedonic depression. Higher scores are indicative of higher levels of anhedonic depression.
Mood and Anxiety Symptom Questionnaire-Anhedonic Depression Subscale | Change from baseline anhedonic depression symptoms (day 1 of study) to 4-weeks post-intervention.
  The Mood and Anxiety Symptom Questionnaire-Anhedonic Depression Subscale (MASQ-AD8) is a self-report assessment used to measure symptoms of anhedonic depression. Higher scores are indicative of higher levels of anhedonic depression.
Ruminative Responses Scale-8 item | Change from baseline rumination levels (day 1 of study) to immediately after the 3-day intervention.
  Ruminative Responses Scale-8 item is commonly used to measure people's general tendency to ruminate. Higher scores suggest higher levels of rumination.
Ruminative Responses Scale-8 item | Change from baseline rumination levels (day 1 of study) to 4-weeks post-intervention.
  Ruminative Responses Scale-8 item is commonly used to measure people's general tendency to ruminate. Higher scores suggest higher levels of rumination.

SECONDARY OUTCOMES:
Mood and Anxiety Symptom Questionnaire-Anxious Arousal Subscale | Change from baseline anxious arousal symptoms (day 1 of study) to immediately after the 3-day intervention.
  Mood and Anxiety Symptom Questionnaire-Anxious Arousal Subscale (MASQ-AA) is a self-report assessment used to measure levels of anxious arousal symptoms. Higher scores on this measure indicate higher levels of anxious arousal.
Mood and Anxiety Symptom Questionnaire-Anxious Arousal Subscale | Change from baseline anxious arousal symptoms (day 1 of study) to 4-weeks post-intervention.
  Mood and Anxiety Symptom Questionnaire-Anxious Arousal Subscale (MASQ-AA) is a self-report assessment used to measure levels of anxious arousal symptoms. Higher scores on this measure indicate higher levels of anxious arousal.
Penn State Worry Questionnaire | Change from baseline anxious apprehension symptoms (day 1 of study) to immediately after the 3-day intervention.
  Penn State Worry Questionnaire is a self-report assessment used to measure symptoms of anxious apprehension. Higher scores on this measure indicate higher levels of anxious apprehension or worry.
Penn State Worry Questionnaire | Change from baseline anxious apprehension symptoms (day 1 of study) to 4-weeks post-intervention.
  Penn State Worry Questionnaire is a self-report assessment used to measure symptoms of anxious apprehension. Higher scores on this measure indicate higher levels of anxious apprehension or worry.
Cognitive and Affective Mindfulness Scale- Revised | Change from baseline mindfulness levels (day 1 of study) to immediately after the 3-day intervention.
  Cognitive and Affective Mindfulness Scale- Revised is a self-report assessment that measures levels of mindfulness. Higher scores on this measure indicate higher levels of mindfulness.
Cognitive and Affective Mindfulness Scale- Revised | Change from baseline mindfulness levels (day 1 of study) to 4-weeks post-intervention.
  Cognitive and Affective Mindfulness Scale- Revised is a self-report assessment that measures levels of mindfulness. Higher scores on this measure indicate higher levels of mindfulness.
Five Facet Mindfulness Questionnaire | Change from baseline mindfulness levels (day 1 of study) to immediately after the 3-day intervention.
  Five Facet Mindfulness Questionnaire is a self-report assessment that measures levels of mindfulness. Higher scores on this measure indicate higher levels of mindfulness.
Five Facet Mindfulness Questionnaire | Change from baseline mindfulness levels (day 1 of study) to 4-weeks post-intervention.
  Five Facet Mindfulness Questionnaire is a self-report assessment that measures levels of mindfulness. Higher scores on this measure indicate higher levels of mindfulness.

CONTACTS AND LOCATIONS:
Overall Officials: Bridget R. Kennedy, Principal Investigator — UT Tyler
Locations (1):
- The University of Texas at Tyler, Tyler, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan at this time to share any data with other researchers. In the event that any data were to be shared, it would only be de-identified and we would follow appropriate guidelines as outlined by UT Tyler's IRB.

REFERENCES:
- [Background] Beevers CG, Clasen PC, Enock PM, Schnyer DM. Attention bias modification for major depressive disorder: Effects on attention bias, resting state connectivity, and symptom change. J Abnorm Psychol. 2015 Aug;124(3):463-75. doi: 10.1037/abn0000049. PMID 25894440
- [Background] Bredemeier K, Spielberg JM, Silton RL, Berenbaum H, Heller W, Miller GA. Screening for depressive disorders using the Mood and Anxiety Symptoms Questionnaire Anhedonic Depression Scale: a receiver-operating characteristic analysis. Psychol Assess. 2010 Sep;22(3):702-10. doi: 10.1037/a0019915. PMID 20822283
- [Background] Bo R, Kraft B, Jonassen R, Harmer CJ, Hilland E, Stiles TC, Haaland VO, Aspesletten MEB, Sletvold H, Landro NI. Symptom severity moderates the outcome of attention bias modification for depression: An exploratory study. J Psychiatr Res. 2021 Jun;138:528-534. doi: 10.1016/j.jpsychires.2021.04.027. Epub 2021 May 5. PMID 33984807
- [Background] Conley MI, Dellarco DV, Rubien-Thomas E, Cohen AO, Cervera A, Tottenham N, Casey BJ. The racially diverse affective expression (RADIATE) face stimulus set. Psychiatry Res. 2018 Dec;270:1059-1067. doi: 10.1016/j.psychres.2018.04.066. Epub 2018 May 19. PMID 29910020
- [Background] Creswell JD. Mindfulness Interventions. Annu Rev Psychol. 2017 Jan 3;68:491-516. doi: 10.1146/annurev-psych-042716-051139. Epub 2016 Sep 28. PMID 27687118
- [Background] Farb NA, Anderson AK, Segal ZV. The mindful brain and emotion regulation in mood disorders. Can J Psychiatry. 2012 Feb;57(2):70-7. doi: 10.1177/070674371205700203. PMID 22340146
- [Background] Fodor LA, Georgescu R, Cuijpers P, Szamoskozi S, David D, Furukawa TA, Cristea IA. Efficacy of cognitive bias modification interventions in anxiety and depressive disorders: a systematic review and network meta-analysis. Lancet Psychiatry. 2020 Jun;7(6):506-514. doi: 10.1016/S2215-0366(20)30130-9. Epub 2020 May 20. PMID 32445689
- [Background] Jones EB, Sharpe L. Cognitive bias modification: A review of meta-analyses. J Affect Disord. 2017 Dec 1;223:175-183. doi: 10.1016/j.jad.2017.07.034. Epub 2017 Jul 18. PMID 28759865
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Mennen AC, Norman KA, Turk-Browne NB. Attentional bias in depression: understanding mechanisms to improve training and treatment. Curr Opin Psychol. 2019 Oct;29:266-273. doi: 10.1016/j.copsyc.2019.07.036. Epub 2019 Jul 31. PMID 31521030
- [Background] Segal, Z. V., Williams, J. M. G., & Teasdale, J. D. (2013). Mindfulness-based Cognitive Therapy for Depression, 2nd ed. New York, NY: The Guilford Press.
- [Background] Schumer MC, Lindsay EK, Creswell JD. Brief mindfulness training for negative affectivity: A systematic review and meta-analysis. J Consult Clin Psychol. 2018 Jul;86(7):569-583. doi: 10.1037/ccp0000324. PMID 29939051
- [Background] Watson D, Clark LA, Weber K, Assenheimer JS, Strauss ME, McCormick RA. Testing a tripartite model: II. Exploring the symptom structure of anxiety and depression in student, adult, and patient samples. J Abnorm Psychol. 1995 Feb;104(1):15-25. doi: 10.1037//0021-843x.104.1.15. PMID 7897037
- [Background] Altman EG, Hedeker D, Peterson JL, Davis JM. The Altman Self-Rating Mania Scale. Biol Psychiatry. 1997 Nov 15;42(10):948-55. doi: 10.1016/S0006-3223(96)00548-3. PMID 9359982